CLINICAL TRIAL: NCT05329545
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled, Multicenter Study of Upifitamab Rilsodotin (XMT-1536) as Post-Platinum Maintenance Therapy for Participants With Recurrent, Platinum-Sensitive, Ovarian Cancer (UP-NEXT)
Brief Title: Upifitamab Rilsodotin Maintenance in Platinum-Sensitive Recurrent Ovarian Cancer (UP-NEXT)
Acronym: UP-NEXT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study Terminated by Sponsor
Sponsor: Mersana Therapeutics (Industry)
Collaborators: GOG Foundation (Network); European Network of Gynaecological Oncological Trial Groups (ENGOT) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: XMT-1536-3
Record Dates: First submitted 2022-03-24; First posted 2022-04-15 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: High Grade Serous Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Cancer
Keywords: Ovarian Cancer; Serous; Maintenance; Antibody Drug Conjugate; Recurrent; Platinum-Sensitive; ADC; Fallopian Tube Cancer; Primary Peritoneal Cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Recurrence

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized, placebo controlled (2:1 upifitamab rilsodotin: placebo). Parallel cohorts.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- XMT-1536 (upifitamab rilsodotin) (Experimental): XMT-1536 (upifitamab rilsodotin)
  Interventions: Drug: Upifitimab rilsodotin
- Placebo (Placebo Comparator): Saline placebo will be administered with same schedule and stopping rules as for the assigned interventions in the Experimental Arm.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Upifitimab rilsodotin — Upifitimab rilsodotin will be administered once every four weeks until completion, disease progression, unacceptable toxicity, voluntary discontinuation, or death (approximately up to 18 months).
  Other Names: XMT-1536 Antibody Drug Conjugate
  Arms: XMT-1536 (upifitamab rilsodotin)
Other: Placebo — Placebo controlled arm.
  Arms: Placebo

SUMMARY:
UP-NEXT is a double-blind, randomized, placebo-controlled study of the antibody-drug conjugate (ADC) XMT-1536 (upifitamab rilsodotin) administered as an intravenous infusion once every four weeks in patients with recurrent, platinum-sensitive high-grade serous ovarian cancer (HGSOC), including fallopian tube and primary peritoneal cancer, expressing high levels of NaPi2b.

DETAILED DESCRIPTION:
This is a multi-center randomized study of XMT-1536 (upifitamab rilsodotin) in patients with tumors expressing high levels of NaPi2b, focusing on patients with recurrent, platinum-sensitive high-grade serous ovarian cancer (HGSOC) including fallopian tube and primary peritoneal cancer. The randomized study design is a double-blind, placebo-controlled study, with a randomization ratio of 2:1. All adverse events will be graded according to the National Cancer Institute (NCI) Common Terminology Criteria version (CTCAE v5.0). Participants must have had 4 to 8 cycles of platinum-based chemotherapy in their most recent treatment regimen, including carboplatin or cisplatin ± paclitaxel, docetaxel, pegylated liposomal doxorubicin or gemcitabine in the 2nd-4th line setting for the treatment of platinum-sensitive recurrent disease, with no evidence of disease (NED)/complete response (CR)/partial response (PR)/ or stable disease (SD) as best response.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must have a histological diagnosis of high grade serous ovarian cancer, which includes fallopian tube and primary peritoneal cancer, that is metastatic or recurrent.
2. Participant must have platinum-sensitive recurrent disease, defined as having achieved either a partial or complete response to 4 or more cycles in their penultimate platinum- containing regimen and their disease progressing more than 6 months after completion of the last dose of platinum containing therapy in the penultimate regimen.
3. Participant must have had 4 to 8 cycles of platinum-based chemotherapy in 2nd to 4th line setting in their most recent treatment regimen as defined below:

   1. Platinum-based chemotherapy regimens allowed immediately preceding enrollment to the study: carboplatin or cisplatin ±: paclitaxel, docetaxel, pegylated liposomal doxorubicin or gemcitabine.
   2. Participant must receive first study treatment infusion between 4 and 12 weeks after completing final dose of platinum in the most recent platinum-based regimen.
4. Participant must have had as their best response to last line of treatment one of the following: No Evidence of Disease (NED); Complete Response (CR); Partial Response (PR); OR Stable Disease (SD)
5. Participants with NED, CR, or PR as their best response to most recent line of treatment and who have not received treatment with a prior PARP inhibitor must have definitive BRCA1 and BRCA2 testing results that demonstrate no evidence of a deleterious BRCA1 or BRCA2 mutation. Somatic BRCA mutation testing is required for participants who are classified as not having a deleterious mutation by germline testing alone.
6. Participant must provide either a tumor tissue block or fresh cut slides for measurement of NaPi2b expression by a central laboratory. If sufficient archival tumor tissue is not available, then a tumor tissue block or slides must be obtained from a fresh biopsy and provided to the central laboratory. Confirmation of a NaPi2b-H/positive tumor by the central laboratory is required prior to randomization.

Exclusion Criteria:

1. Participant has received prior treatment with mirvetuximab soravtansine or another ADC containing an auristatin or maytansinoid payload.
2. Participant has received bevacizumab in combination with last platinum-based regiment or plans to receive maintenance therapy outside the study intervention.
3. Participant has clinical signs or symptoms of gastrointestinal obstruction and/or requirement for parenteral hydration or nutrition.
4. Participant has ascites or pleural effusion managed with therapeutic paracentesis or thoracentesis within 28 days prior to signing the principal study consent form.
5. Participant has history of cirrhosis, hepatic fibrosis, esophageal or gastric varices, or other clinically significant liver disease. Testing beyond laboratory studies otherwise defined in the eligibility criteria, to diagnose potentially clinically significant liver disease based on risk factors such as hepatic steatosis or history of excessive alcohol intake, will be based on clinical judgement of the investigator.
6. Participant has history of or suspected pneumonitis or interstitial lung disease.
7. Participant has untreated CNS metastases (including new and progressive brain metastases), history of leptomeningeal metastasis, or carcinomatous meningitis.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2022-06-23 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-09-29 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) assessed by Blinded Independent Central Review (BICR) using Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 | Up to 12 months after the last dose for the last participant.
  PFS is defined as the time from randomization to the earliest date of progressive disease as assessed by BICR per RECIST Version 1.1 or death due to any cause.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to an average of 4 years. Follow up assessments for survival data will continue every 90 days following completion of treatment.
  OS is defined as the time from randomization to the date of death due to any cause.
Progression-free Survival (PFS) as assessed by Investigator using Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 | Up to 12 months after the last dose for the last participant.
  PFS is defined as the time from randomization to the earliest date of progressive disease as assessed by Investigator per RECIST Version 1.1 or death due to any cause.
Adverse events (AEs) based on NCI CTCAE Version 5.0 | Up to 60 days past last dose
  Incidence and toxicity grade of AEs.
Changes in Eastern Cooperative Oncology Group (ECOG) performance status | Up to 60 days past last dose.
  Assessment of ECOG performance status using ECOG performance scale.
Objective Response Rate (ORR) as assessed by Investigator using RECIST Version 1.1 | Up to 12 months after the last dose for the last participant.
  ORR is the percentage of patients achieving a confirmed complete response (CR) or partial response (PR) as assessed by Investigator per RECIST Version 1.1.
Number of participants using concomitant medications | Up to 60 days past last dose.
  Assessment of concomitant medication usage.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Burger, MD, Study Director — Mersana Therapeutics
Locations (30):
- United States (28):
  - HonorHealth Research Institute - HonorHealth VGPCC Biltmore, Phoenix, Arizona
  - The University of Arizona Cancer Center, Tucson, Arizona
  - University of California Los Angeles, Gynecologic Oncology Clinic, Los Angeles, California
  - University of California, Irvine Medical Center, Orange, California
  - Sarasota Memorial Hospital, Sarasota, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - WK Physicians, Shreveport, Louisiana
  - Karmanos Cancer Institute - Detroit, Detroit, Michigan
  - Billings Clinic, Billings, Montana
  - Methodist Hospital, Omaha, Nebraska
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Center of Hope, Reno, Nevada
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Southwest Women's Oncology, Albuquerque, New Mexico
  - University Hospitals Cleveland Medical Center, Seidman Cancer Center, Cleveland, Ohio
  - Kettering Health Cancer Center, Kettering, Ohio
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Willamette Valley Cancer Institute and Research Center, Eugene, Oregon
  - Legacy Good Samaritan Medical Center - Legacy Medical Group - Gynecologic Oncology, Portland, Oregon
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Sanford Gynecologic Oncology, Sioux Falls, South Dakota
  - Avera McKennan d/b/a Avera Research Institute, Sioux Falls, South Dakota
  - Texas Oncology P.A. - Austin, Austin, Texas
  - Texas Oncology - DFWW, Bedford, Texas
  - Texas Oncology - Tyler, Tyler, Texas
  - VCU Massey Cancer Center, Richmond, Virginia
  - University of Wisconsin Clinical Science Center, Madison, Wisconsin
  - Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin
- Epworth Richmond, Richmond, Victoria, Australia
- Sherbrooke University Hospital Centre, Québec, Sherbrooke, Canada

IPD SHARING:
Plan to Share IPD: No